CLINICAL TRIAL: NCT02643186
Title: Vaginal Misoprostol Versus Bilateral Uterine Artery Ligation in Decreasing Blood Loss in Trans-abdominal Myomectomy , a Randomized Control Trail
Brief Title: Vaginal Misoprostol Versus Bilateral Uterine Artery Ligation in Decreasing Blood Loss in Trans-abdominal Myomectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, aliaa mohamed ali, university, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ASUMH
Record Dates: First submitted 2015-12-21; First posted 2015-12-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Vaginal Misoprostol and Bilateral Uterine Artery Ligation in Decreasing Blood Loss in Trans-abdominal Myomectomy
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- misoprostol group (Active Comparator): preoperative vaginal misoprostol in decreasing blood loss in transabdominal myomectomy
  Interventions: Drug: preoperative vaginal misoprostol
- uterine artery ligation group (Active Comparator): bilateral uterine artery ligation in decreasing blood loss in transabdominal myomectomy
  Interventions: Procedure: bilateral uterine artery ligation

INTERVENTIONS:
Drug: preoperative vaginal misoprostol — preoperative vaginal misoprostol 400 micrograms 1 hour before surgery
  Other Names: cytotec
  Arms: misoprostol group
Procedure: bilateral uterine artery ligation — bilateral ascending uterine artery ligation at the level of uterine isthmus with 2/0 vicryl sutures
  Other Names: devascularization
  Arms: uterine artery ligation group

SUMMARY:
The study aims at comparison between the effect of preoperative misoprostol and bilateral uterine artery ligation regarding their effect to decrease blood loss in transabdominal myomectomy.

ELIGIBILITY:
Inclusion Criteria:

* women in the reproductive age (20-40 years) diagnosed as having uterine fibroids who are consenting to have trans- abdominal myomectomy in the postmenstrual period diagnosed by: clinical symptoms and signs:
* abnormal uterine bleeding (menorrhagia or/and metrorrhagia)
* pain (dull aching lower abdominal pain or dysmenorrhea)
* pressure symptoms (dyspareunia, dysuria, dyschezia or /and backache)
* progressive abdominal enlargement (abdominal swelling) ultrasound (abdominal or transvaginal) to confirm the clinical diagnosis:
* maximum diameter of the largest fibroid is greater than 4 cm
* maximum number of uterine myomas is not to be more than 5 myomas
* uterine fibroid may be subserous or intramural

Exclusion Criteria:

* obesity (BMI >30 kg/m2)
* cardiac, endocrine, pulmonary or hematological disease (including anemia; hemoglobin level below 10 gm/dl)
* patients known to be allergic to prostaglandin preparations
* patients who received preoperative hormonal therapy (GnRH analogue)
* patients presented by or with suspected malignant gynecological disease patients diagnosed as having submucous uterine fibroids, cervical or supracervical fibroids, broad ligamentary fibroids and pedunculated fibroids patients with contraindication to general anaesthesia
* patients with positive pregnancy test
* virgin patients

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
estimated intraoperative blood loss measured in milliliters | 60 min

SECONDARY OUTCOMES:
the need of intra-operative blood transfusion | 60 min
  Below a hemoglobin concentration of 7 g/dL requiring blood transfusion. It is indicated when intra-operative blood loss exceeds 15% of the patient's estimated blood volume, which is equal to the patient's weight in kilograms multiplied by 10).
the need for conversion from myomectomy to hysterectomy | 60 min
  It is indicated when there is uncontrolled intra-operative hemorrhage affecting the patient's vital signs and not responsive to conservative measures when it is impossible to reconstruct the uterus because of the many defects left by the removal of multiple fibroids
operative time in minutes | 60 min
intraoperative or postoperative complications | 24 hours
differance between pre and post operative hemoglobin and hematocrit levels | 24 hours
duration of hospital stay in days | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt